CLINICAL TRIAL: NCT04977596
Title: Grade 3 Pancreatic Neuroendocrine Tumors on MDCT: Establishing a Diagnostic Model and Comparing Survival Against Pancreatic Ductal Adenocarcinoma
Brief Title: Related Studies of Imaging Features and Prognosis Between Pancreatic Neuroendocrine Tumors and Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other); The First Affiliated Hospital of the Fourth Military Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: yurisheng
Record Dates: First submitted 2021-07-12; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2020-03

CONDITIONS: Neuroendocrine Tumor of Pancreas; Carcinoma, Pancreatic; CT
MeSH Terms: conditions — Adenoma, Islet Cell; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group PNETs: The investigators retrospectively analyzed data for patients who underwent contrast-enhanced MDCT for the evaluation of G3 PNETs at the Second Affiliated Hospital of Zhejiang University School of Medicine (n = 12) between January 2011 and May 2019, patients with G3 PNET who underwent MDCT at the First Affiliated Hospital of Zhejiang University School of Medicine (n = 4) and the Military Medical University of Air Force (The Fourth Military Medical University) (n = 4) between January 2013 and October 2018
  Interventions: Other: No intervention
- Group PDAC: Patients with PDAC who underwent MDCT at the Second Affiliated Hospital of Zhejiang University School of Medicine (n = 58) from February 2014 to August 2015.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Retrospective study without intervention

SUMMARY:
1. Imaging findings (including CT and MRI images) of both well-differentiated G3 PNET and poorly differentiated PNET were studied;
2. The CT imaging findings of G3 stage PNET and pancreatic cancer were compared to establish a Logistic regression diagnostic model, and the survival analysis of the two was compared.
3. Cox regression was used to study the risk factors for survival prognosis of well-differentiated and poorly differentiated PNET based on CT image features

DETAILED DESCRIPTION:
According to the latest WHO Classification of Neuroendocrine Neoplasms (NET) in 2019, pancreatic neuroendocrine neoplasms (PNET) are divided into well-differentiated and poorly differentiated PNETs.The former is divided into G1, G2, and well differentiated G3.There are few studies on the survival outcomes of these two differentiated PNET types.The G3 imaging manifestations of the two types of differentiation have not been studied yet, and G3 PNET is often clinically misdiagnosed as pancreatic cancer, so it is necessary to differentiate the imaging manifestations and survival time of the two types.

A total of 71 patients with PNET in our hospital from January 2012 to January 2019 and 58 patients with pancreatic cancer from February 2014 to August 2015 were retrospectively collected. Complete survival time data of all patients after telephone follow-up were obtained.Since G3 PNET is very rare, the investigators enrolled 9 patients with G3 PNET in the First Affiliated Hospital of Zhejiang University School of Medicine and 7 patients with G3 PNET in the Affiliated Hospital of Air Force Military Medical University from January 2013 to October 2018.

CT images of PNET and pancreatic cancer were analyzed independently by two radiologists specializing in abdominal diagnosis, in which G3 lesions were evaluated simultaneously on MRI images and the others were evaluated only on CT images.Records clinical data and imaging characteristics: gender, age, tumor markers, tumor shape, size, tumor characteristics, edge, the expansion of the shrinking, pancreas, pancreatic pancreatitis, enhancement scan, arterial phase and portal phase lesions and the ratio of pancreatic parenchyma around, liver metastasis, peripheral vascular invasion, lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis by pathology and detailed pathological information
2. Enhanced CT examination or biopsy were performed within 2 months before surgery
3. There was no preoperative radiotherapy or chemotherapy

Exclusion Criteria:

1. No Ki-67 index
2. CT value cannot be measured by ROI because of pancreatic atrophy and other reasons
3. No enhanced images or missing images

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators retrospectively analyzed data for patients who underwent contrast-enhanced MDCT for the evaluation of G3 PNETs at the Second Affiliated Hospital of Zhejiang University School of Medicine (n = 12) between January 2011 and May 2019, patients with G3 PNET who underwent MDCT at the First Affiliated Hospital of Zhejiang University School of Medicine (n = 4) and the Military Medical University of Air Force (The Fourth Military Medical University) (n = 4) between January 2013 and October 2018, and consecutive patients with PDAC who underwent MDCT at the Second Affiliated Hospital of Zhejiang University School of Medicine (n = 58) from February 2014 to August 2015.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Tumor size | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  Maximum surface size of the lesion (cm)
Tumor location | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  Locations of the pancreas: head, neck, body and tail
Number of lesions | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  Number of lesions
Margin | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  well-defined or ill-defined
tumor texture | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  solid；solid and cystic；complex cystic
Pancreatic tail contraction | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  yes or no
Complicated pancreatitis | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  yes or no
Pancreatic duct/bile duct dilatation | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  yes or no
Extrapancreatic tissue invasion | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  yes or no
Hepatic metastasis | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  yes or no
Lymphatic metastasis | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  yes or no
CT value of pancreas plain scan | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  CT value of pancreas plain scan
CT value of lesion plain scan | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  CT value of lesion plain scan
CT value of pancreas artery phase | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  CT value of pancreas artery phase
CT value of lesion artery phase | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  CT value of lesion artery phase
CT value of pancreas portal phase | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  CT value of pancreas portal phase
CT value of lesion portal phase | preoperative contrast-enhanced CT performed within 2 months before surgery or biopsy
  CT value of lesion portal phase

CONTACTS AND LOCATIONS:
Overall Officials: Risheng Yu, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No